CLINICAL TRIAL: NCT04190992
Title: The Effect of E-Based Technology to Provide Personalized Decision Aid on Breast Reconstruction for Women With Breast Cancer
Brief Title: E-Based Technology to Provide Decision Aid on Breast Reconstruction for Women With Breast Cance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Su-Ying Fang, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B-ER-106-072
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Decision Support Technique; Breast Cancer
Keywords: Decision aid; Breast reconstruction; E-based Technology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application (APP) group (Experimental): After completing the questionnaires at baseline, participants in the experimental group will be asked to receive a pamphlet and an E-based & personalized breast reconstruction surgery decision aid at clinic.
  Interventions: Other: E-based & personalized breast reconstruction surgery decision aid; Other: Usual care
- Usual care group (Other): After completing the questionnaires at baseline, participants in the control group will only receive a pamphlet as usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: E-based & personalized breast reconstruction surgery decision aid — This decision aid contains information regarding surgical options, including breast reconstruction and mastectomy, such as the advantages and disadvantages, the complication probabilities of each option, a value clarification exercise for the patient's self-evaluation, and a summary of the participant's decision-making process.
  Other Names: APP decision aid
  Arms: Application (APP) group
Other: Usual care — A pamphlet introduce the introduction of types of surgery

SUMMARY:
Using decision aids has been demonstrated to support women to make treatment decision effectively. However, these studies focused on the decision of receiving breast conservative surgery or mastectomy, had short term follow-ups on decision satisfaction.The aims of this study were: Evaluate the effect of E-based & personalized breast reconstruction surgery decision aid on women's decision satisfaction and mental health.

DETAILED DESCRIPTION:
Randomized controlled trial will be used to examine the effect of E-based & personalized breast reconstruction surgery decision aid on decision satisfaction, body image, anxiety and depression. Participants will be randomly assigned into either experimental or control groups with 88 women in each group. After completing the questionnaires at baseline, participants in the experimental group will be asked to receive a E-based & personalized breast reconstruction surgery decision aid at clinic. Control group will only receive pamphlet and usual care. All participants will be followed up 1 week after consultation, and 1 month, 8 month and 12 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 20 years or under 20 years but married
* females newly diagnosed with breast cancer who are candidates for mastectomy
* ability to read and speak Taiwanese or Mandarin

Exclusion Criteria:

* Women with cancer recurrence
* poor cognitive function
* diagnosed with psychiatric disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Body image | Pre-surgery, 1 month, 8 month, 12 month post surgery
  The Body Image Scale (BIS) has ten items rated on a four-point Likert scale (0 [not at all] to 3 [very much]), with total scores ranging from 0 to 30. Higher scores indicate greater BI distress.
Decision Regret | 1 month, 8 month, 12 month post surgery
  Decision Regret Scale (DRS) accesses "distress or remorse after a surgery decision". This instrument contains 5 items. The items were summed, divided by 5, and multiplied by 25. Higher scores indicate greater decision regret.
Decision conflict | Pre-surgery, 1 week after intervention
  Decision Conflict Scale (DCS) accesses the perception of uncertainty in information, values or support for surgery options. This instrument contains 16 items and was developed by O'Connor. The items were summed, divided by 16, and multiplied by 25. Higher scores indicate greater decision conflict.

SECONDARY OUTCOMES:
Anxiety | Pre-surgery, 1 month, 8 month, 12 month post surgery
  The Hospital Anxiety and Depression Scale (HADS) assesses symptoms of anxiety and depression. The HADS includes 14 items, of which 7 measure anxiety, and 7 measure depression. All items are scored using a 0-3 point scale, with higher scores indicating more depressive symptoms. Cut-off scores are used to categorize anxiety and depressive symptoms, with values of over 8 indicating possible anxiety and depression, and 11 or above indicating probable anxiety.
Depression | Pre-surgery, 1 month, 8 month, 12 month post surgery
  The Hospital Anxiety and Depression Scale (HADS) assesses symptoms of anxiety and depression. The HADS includes 14 items, of which 7 measure anxiety, and 7 measure depression. All items are scored using a 0-3 point scale, with higher scores indicating more depressive symptoms. Cut-off scores are used to categorize anxiety and depressive symptoms, with values of over 8 indicating possible anxiety and depression, and 11 or above indicating probable depression.
Involvement in the Breast Reconstruction (BR) decision-making process scale | 1 week after intervention
  Involvement in the BR decision-making process was divided into two subscales, one accesses the perception of medical information about surgery obtained with 6 items and the other assesses the perception of partners' involvement in the BR decision-making process with 7 items. The scale used a five-point Likert scale (1 [strongly disagree] to 5 [strongly agree]); the higher the score, the greater the amount of information the participants believed they had obtained and the greater the participants perceived their partner's involvement in the BR decision-making process.

CONTACTS AND LOCATIONS:
Overall Officials: Su-Ying Fang, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Fang SY, Lin PJ, Kuo YL. Long-Term Effectiveness of a Decision Support App (Pink Journey) for Women Considering Breast Reconstruction Surgery: Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 10;9(12):e31092. doi: 10.2196/31092. PMID 34890354